CLINICAL TRIAL: NCT00864240
Title: Dose Response of Clobex 0.05% Lotion
Brief Title: The Dose-response "Pilot" Study of Topically Delivered Clobetasol Propionate Lotion in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Christine Winslow, Director of Clinical Development, Actavis Inc
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10504909
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Healthy
Keywords: Vasoconstriction; Clobetasol; Healthy adult females
MeSH Terms: interventions — Clobetasol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Clobex TM 0.05% Lotion, single exposure
  Interventions: Drug: Clobex TM (Clobetasol) 0.05% Lotion, single exposure

INTERVENTIONS:
Drug: Clobex TM (Clobetasol) 0.05% Lotion, single exposure — Subjects received Galderma Laboratories, L.P. formulated products
  Other Names: Clobetasol

SUMMARY:
To determine the dose-response relationship for Clobex TM (clobetasol propionate) Lotion, 0.05%. This information will be used to estimate the ED50, D1, D2 parameters for use in a full bioequivalence study.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Randomized, open label, one period, dose response, vasoconstrictor assay study.

Official Title: Dose Response of Clobex 0.05% Lotion

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

· Vasoconstrictor Response

ELIGIBILITY:
Inclusion Criteria:

* Non-tobacco-using female subjects, 18 to 50 years of age, inclusive.
* A demonstrated blanching response to Clobex TM (clobetasol propionate) Lotion, 0.05 %.
* A body mass index (BMI) 30 kg/m2 or less as calculated according to Novum Standard Operating Procedures.
* Good health as determined by lack of clinically significant abnormalities in medical history and clinical assessment, as judged by the Investigator.
* Signed and dated informed consent form which meets all criteria of current FDA regulations.

Exclusion Criteria:

* History of allergy to any systemic or topical corticosteroid (including clobetasol) or to any cream, lotion, ointment, gel, cotton, soap, cosmetic, rubber, or tape, which in the opinion of the Investigator would compromise the safety of the subject or the study.
* Presence of any skin condition or coloration that would interfere with placement of test sites or the response or assessment of skin blanching.
* Significant history or current evidence of chronic infectious disease, system disorder (especially hypertension or circulatory disease), or organ dysfunction.
* Presence of a medical condition requiring regular treatment with prescription drugs.
* Drug or alcohol addiction requiring treatment (in-patient or out-patient) in the 12 months prior to dosing.
* Use of any topical dermatological drug therapy (including topical corticosteroids) on the flexor surface of the ventral forearms in the 30 days prior to dosing.
* Use of any tobacco products in the 30 days prior to dosing.
* Receipt of any drug as part of a research study within 30 days prior to initial study dosing.
* Pregnant or lactating.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-10; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Vasoconstriction response | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Soran Hong,, M.D., Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Houston, Texas, United States